CLINICAL TRIAL: NCT03865797
Title: Effectiveness of Core Work and Sports Bandage to Improve Ankle Instability in Rugby Players: A Pilot Study
Brief Title: Core Work and Sports Bandage in Rugby Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AZul
Record Dates: First submitted 2019-03-04; First posted 2019-03-07 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Rugby

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Before carrying out each session of the intervention, each subject included in the experimental group will have a sports bandage on both ankles. The intervention by motor control will consist of the application of a series of Core exercises. The exercises will be carried out with the subjects in different positions of prone, lateral and supine position, for the Core musculature. The exercises will be repeated 10 times each and there will be 8 different exercises: roll up, mermaid, raised crossed, stretch two leg back, shoulder bridge and leg pull up. The duration of each session will be 15 minutes, with two sessions per week, during a period of 4 weeks.
  Interventions: Other: Experimental
- Control (Active Comparator): The intervention by motor control will consist of the application of a series of Core exercises. The exercises will be carried out with the subjects in different positions of prone, lateral and supine position, for the Core musculature. The exercises will be repeated 10 times each and there will be 8 different exercises: roll up, mermaid, raised crossed, stretch two leg back, shoulder bridge and leg pull up. The duration of each session will be 15 minutes, with two sessions per week, during a period of 4 weeks.
  Interventions: Other: Control active

INTERVENTIONS:
Other: Experimental — Each session will last approximately 15 minutes, taking place during 2 days a week, in a period of 4 weeks. The intervention will be done before the training session. The intervention by motor control will consist of the application of a series of Core exercises. The exercises will be carried out with the subjects in different positions of prone, lateral and supine position, for the Core musculature. The exercises will be repeated 10 times each and there will be 8 different exercises: roll up, mermaid, raised crossed, stretch two leg back, shoulder bridge and leg pull up.The intervention will be done before the training session.
  Other Names: Ankle stability
  Arms: Experimental
Other: Control active — Each session will last approximately 15 minutes, taking place during 2 days a week, in a period of 4 weeks. The intervention will be done before the training session. The intervention by motor control will consist of the application of a series of Core exercises. The objective of the application of these exercises is to increase the control of the Core, and therefore improve the stability both central and of members. The exercises will be carried out with the subjects in different positions of prone, lateral and supine position, for the Core musculature. The exercises (13) will be repeated 10 times each and there will be 8 different exercises: roll up, mermaid, raised crossed, stretch two leg back, shoulder bridge and leg pull up.
  Other Names: Ankle stability
  Arms: Control

SUMMARY:
Introduction. Lower limb injuries are characteristic of rugby players. Core exercises aim to improve ankle stability. The ankle bandage in 8 is used in the approach to injuries to provide better stability in the joint.

Objectives. To assess the effectiveness of an intervention through motor control and bandage on lower limb stability in rugby players from 18 to 40 years old.

Study design. Randomized, single-blind clinical study with a follow-up period. Methodology. Twenty-five rugby players will be recruited to be randomized to the two study groups: experimental (specific exercises for the Core area and ankle bandage) and control (Core motor control). The intervention will last 4 weeks, with 2 weekly sessions of 15min each. The study variables will be: core motor control (measured with plate test, trunk flexion test and modified Biering-Sorensen test) and the stability of the lower limbs (measured with Double Heel Rise and Single Heel Rise test). A descriptive analysis will be carried out calculating the main statistical characteristics. Through an analysis of Shapiro-Wills the normality of the study groups will be calculated, and through an analysis with the parametric tests of t-student and ANOVA of repeated measures, we will evaluate the difference after the evaluations in both groups and the intra-e intersubject, respectively.

Expected results. Increased motor control of the core and stability of lower limbs.

ELIGIBILITY:
Inclusion Criteria:

* Rugby players
* Both gender
* From 18 to 40 years old
* Federated.

Exclusion Criteria:

* At the time of the study, they present an injury that prevents them from carrying out the proposed intervention
* Included in a personal training regime
* With musculoskeletal injuries in the ankle in the last 3 months
* Not sign the informed consent document.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2019-04-10 (Actual); Study Completion 2019-06-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline central stability after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The assessment of the central stability will be carried out with the modified Biering-Sorensen test. The subject must remain prone on a stretcher, while the part of the trunk should protrude through the front of the stretcher and completely parallel to the floor. The arms will remain crossed on the chest touching the shoulders at all times. The test ends when the subject supports any part of his body on the floor. The normative values of this test are 146 seconds for men and 189 for women, with the second being the unit of measurement for this test.

SECONDARY OUTCOMES:
Change from baseline Core rating after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  By means of the lateral plate test, which is a test adapted from the exercise of the side plate, we will evaluate the Core. The subject will be placed in lateral decubitus with the elbow resting on the floor, asking him to raise the hip and remain static for the established time. The most characteristic modification is the crossing of the arm in front of the trunk to touch the shoulder of the arm that is in contact with the ground. The unit of measurement is of time (in seconds). The normative values of lumbopelvic stability in men range from 94 to 97 seconds, being in women from 72 to 77 seconds.
Change from baseline trunk strength after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  By means of the isometric trunk flexion test the trunk force will be measured in a situation similar to the sit up, but without movement. The subject will be placed in the supine position, with the knees bent and feet grasped by the assessor or by straps, but with a trunk flexion at 60 degrees (a square can be used for its concretion). The test will end when this angle varies, with the unit of measurement being the second. The normative value range is 149 to 144 seconds.
Change from baseline ankle stability after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The stability of the ankle will be measured with the Double Heel Rise test, which consists of asking the athlete to stand on tiptoe with both feet at the same time and the evaluator will measure the calcaneus of the foot. If, on tiptoe, the calcaneus does not change its position from valgus to varus (rearward projection to supinated hindfoot), it means that the posterior tibial muscle is not in good condition. However, when the player's heel changes its position from valgus to varus, the test will be negative and the posterior tibial will be in good condition.
Change from baseline ankle stability after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The stability of the ankle will be measured with the Single Heel Rise test, which consists in requesting the athlete to stand on tiptoe only with the foot to be evaluated, while the evaluator will measure the calcaneus bone of the foot. If, on tiptoe, the calcaneus does not change its position from valgus to varus (rear right to backward supinated), it means that the posterior tibial muscle of that leg is not in good condition. However, when the player's heel changes its position from valgus to varus, the test will be negative and the posterior tibial will be in good condition.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Europea de Madrid, Madrid, Comunity of Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided